CLINICAL TRIAL: NCT06556407
Title: Effect of Renal Denervation on Blood Pressure in Patients With Treatment Resistant Hypertension, End-stage Chronic Kidney Disease and Hemodialysis
Brief Title: Effect of Renal Denervation on Bood Pressure in Patients on Hemodialysis
Acronym: RDN-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-388-MDz
Record Dates: First submitted 2024-08-05; First posted 2024-08-16 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Treatment Resistant Hypertension; Chronic Hemodialysis

STUDY DESIGN:
Intervention Model Description: prospective, single-center feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Other): Intervention: Renal denervation
  Interventions: Device: renal denervation

INTERVENTIONS:
Device: renal denervation — ultrasound based renal denervation

SUMMARY:
The RDN-HD Study is a prospective, single-center feasibility study. All patients included will undergo endovascular ultrasound-based RDN (no sham group, no blinding). The purpose of the RDN-HD Study is to demonstrate that ultrasound-based RDN is safe in patients with TRH and ESRD hemodialysis and reduces 24-h ambulatory BP.

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) and hemodialysis have a very high risk for cardiovascular events and a very high cardiovascular mortality. Uncontrolled treatment resistant hypertension (TRH) is an important factor driving this very high cardiovascular event risk. Clinical and experimental studies have clearly shown that sympathetic nerve activity is increased in patients with chronic kidney disease (CKD) and substantially aggravates the progression of CKD. In patients with ESRD and chronic hemodialysis bilateral nephrectomy reduced increased sympathetic nerve activity. Interestingly, kidney transplantation did not normalize peripheral sympathetic activity unless the native kidneys were removed. Thus, afferent sensory nerve signaling from the diseased kidneys to the central nervous system is an important pathophysiologic mechanism in CKD leading to sympathetic overactivity and hypertension. Clinical studies have demonstrated that invasive, catheter-based renal denervation (RDN) decreases the sympathetic nerve activity in the whole body and in particular in the kidneys

ELIGIBILITY:
Inclusion Criteria:

* Uncontrolled treatment resistant hypertension (despite intake of 3 different classes of antihypertensive medications) confirmed by 24-h ambulatory blood pressure according to current guidelines (ESH 2023) (office blood pressure ≥ 140/ and/ or ≥ 90 mmHg and ambulatory blood pressure ≥ 130/ and/or ≥ 80 mmHg
* end-stage renal disease on chronic hemodialysis
* Stable hemodialysis regime for at least 3 months based on the decision of the treating physician
* Patient is adhering to a stable drug regimen without changes for a minimum of 4 weeks.
* Individual is ≥ 18 years of age, male and female patients are included.

Exclusion Criteria:

* Episodes of sustained systolic and/or diastolic hypotension according to 24-h ambulatory blood pressure or dialysis protocols which in the eyes of the treating physician would interfere with a safe renal denervation treatment of the patient
* Known hemodynamically or anatomically significant renal artery abnormality or stenosis in either renal artery which in the eyes of the interventionalist would interfere with safe catheter placement
* Prior renal denervation procedure
* Anatomic or functional solitary kidney, kidney transplantation
* Severe atherosclerotic disease or artery calcification preventing the assessment of reliable BP measurements
* Endocrine hypertension other than obstructive sleep apnea
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 3 months of the screening visit
* Acute episode of systemic and renal disease requiring uptitration of any immunosuppressive drug regimen within the last 3 months
* Subject is pregnant, nursing, or intends to become pregnant
* Enrollment in another interventional research protocol.
* Any condition that, at the discretion of the investigator, would preclude participation in the study (e.g. non-adherence)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints and adverse effects | during 6 months post-procedure
  A major combined safety endpoint is the incidence of any major adverse events (MAE) through the 6 months FU
Change in 24-h ambulatory systolic blood pressure between baseline and 3 months post-procedure | baseline and 3 months post-procedure

SECONDARY OUTCOMES:
Change in 24-h ambulatory systolic blood pressure between baseline and 6 months post-procedure | between baseline and 6 months post-procedure.
Change in 24-h ambulatory diastolic blood pressure between baseline and 3, 6 months post-procedure | baseline and 3, 6 months post-procedure.
Change in office (attended) systolic and diastolic blood pressure between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure
Change in systolic and diastolic home blood pressure between baseline and 3, 6 months post-procedure. | between baseline and 3, 6 months post-procedure
Number of antihypertensive drugs, doses, classes at 3, 6 months post-procedure compared to baseline. | at 3, 6 months post-procedure compared to baseline.
Change in bio-impedance parameters between baseline and 3, 6 months post-procedure to assess the volume status. | between baseline and 3, 6 months post-procedure
Change in central systolic and diastolic blood pressure, central pulse pressure and pulse wave velocity between baseline and 3,6 months post procedure | between baseline and 3,6 months post procedure
Change in retinal arteriolar wall to lumen ratio between baseline and 3,6 months post procedure | between baseline and 3,6 months post procedure
Change in average daytime/night-time ambulatory systolic blood pressure between baseline and 3, 6 months post-procedure. | between baseline and 3, 6 months post-procedure.
Change in average daytime/night-time ambulatory diastolic blood pressure between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure
Change in office (attended) and ambulatory heart rate between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure
Changes in dipper/non-dipper patterns between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure
Change in retinal arterial remodeling between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure
Change in retinal capillary density between baseline and 3, 6 months post-procedure | between baseline and 3, 6 months post-procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich Alexander University Erlangen Nuremberg, Department of Nephrology and Hypertension, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No